CLINICAL TRIAL: NCT02678182
Title: Planning Treatment for Oesophago-gastric Cancer: a Randomised Maintenance Therapy Trial
Brief Title: Planning Treatment for Oesophago-gastric Cancer: a Maintenance Therapy Trial
Acronym: PLATFORM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: MedImmune LLC (Industry); Clovis Oncology, Inc. (Industry); Eli Lilly and Company (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3804
Record Dates: First submitted 2015-02-13; First posted 2016-02-09 (Estimated); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Adenocarcinoma of the Oesophagus; Adenocarcinoma of the Gastro-oesophageal Junction; Adenocarcinoma of the Stomach
MeSH Terms: interventions — Capecitabine; durvalumab; Trastuzumab; rucaparib; Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A1: Surveillance (No Intervention): Patients in this Arm will follow current UK standard of care for this setting and will be reviewed every 4 weeks
- Arm A2: Capecitabine Maintenance (Experimental): 1250 mg/M2/DAY on days 1-21
  Interventions: Drug: Capecitabine
- Arm A3: MEDI4736 (Durvalumab) (Experimental): IV treatment on day 1 +15, on a 28 day cycle.
  Interventions: Drug: MEDI4736 (Durvalumab)
- Arm B1: Trastuzumab Maintenance (Active Comparator): 6mg/kg on day 1 every 21 days
  Interventions: Drug: Trastuzumab
- Arm A4: Rucaparib (Experimental): 600mg PO twice daily
  Interventions: Drug: Rucaparib
- Arm A5: Capecitabine and Ramucirumab (Experimental): capecitabine 1250 mg/m2/day PO in two divided doses continuously from days 1-21 of each 21 day cycle (see section 12) and ramucirumab 8mg/kg IV day 1 and day 8
  Interventions: Drug: Capecitabine; Drug: Ramucirumab

INTERVENTIONS:
Drug: Capecitabine — 1250 mg/m2/day, 21 day cycle
  Arms: Arm A2: Capecitabine Maintenance; Arm A5: Capecitabine and Ramucirumab
Drug: MEDI4736 (Durvalumab) — IV treatment on days 1&15 of 28 day cycle
  Arms: Arm A3: MEDI4736 (Durvalumab)
Drug: Trastuzumab — 6mg/kg on day 1 cycle every 21 days
  Arms: Arm B1: Trastuzumab Maintenance
Drug: Rucaparib — 600mg PO twice daily
  Arms: Arm A4: Rucaparib
Drug: Ramucirumab — ramucirumab 8mg/kg IV day 1 and day 8
  Arms: Arm A5: Capecitabine and Ramucirumab

SUMMARY:
To evaluate the efficacy of maintenance therapies following completion of standard first-line chemotherapy in patients with locally advanced or metastatic HER-2 positive or HER-2 negative oesophago-gastric adenocarcinomas.

DETAILED DESCRIPTION:
This is a prospective, open label, multicentre, randomised phase II clinical trial. An adaptive trial design is proposed to allow ineffective treatments to be discontinued early, and to potentially add novel treatment arms as the trial progresses.

Patients will initially receive standard chemotherapy for their locally advanced or metastatic oesophago-gastric adenocarcinoma, according to local practice based upon their HER-2 status (tested locally). In order to be eligible for trial entry, HER-2 negative patients should have received a platinum-fluoropyrimidine based chemotherapy doublet of either cisplatin + capecitaine (CX), oxaliplatin + capecitabine (CAPOX), or 5FU + oxaliplatin (FOLFOX) (Arm A), whilst HER-2 positive patients (IHC 3+ or IHC 2+ and FISH positive) should have received cisplatin in combination with either capecitabine or 5-FU (CX or CF) plus trastuzumab chemotherapy (Arm B). Potentially eligible patients will be registered with the trials office whilst undergoing first line chemotherapy.

Patients will become eligible for trial recruitment and randomisation after 18 weeks standard chemotherapy with stable disease (SD) or better on the end-of-treatment CT scan. Please note: if your patient has been receiving a regimen delivered every three weeks (e.g. CX) they should have completed 6 cycles. If your patient has been receiving a regimen delivered every 2 weeks (e.g. FOLFOX) they should have received 9 cycles of treatment. Eligible patients will then be randomised according to HER-2 status as follows:

* HER-2 positive patients (~20%) will be assigned maintenance single-agent trastuzumab (current UK standard)
* HER-2 negative patients (~80%) will be randomised 1:1 between surveillance (current UK standard) and maintenance capecitabine.

Patients will be stratified according to: centre region, disease extent and performance status (0 versus 1 versus 2).

Review of patients will occur every 4 weeks in the surveillance arm. In maintenance therapy arms, patients will be reviewed every 3 or every 4 weeks depending upon the treatment strategy. CT assessments of response will occur every 12 weeks (3 months) in all arms of the trial. Treatment will be continued until disease progression, unacceptable toxicity, or patient withdrawal for another reason.

The trial is being run from the RM GI and Lymphoma CTU with Professor David Cunningham as the Chief Investigator (CI). Effective arms in the phase II portion of the trial may be taken forward into a phase III maintenance trial powered for overall survival. It is also hoped that, as more robust data becomes available for other biomarker-selected populations (e.g. MET-positive, FGFR-amplified), it may be possible to amend the overall trial design to incorporate these biomarker-targeted maintenance therapies in the HER-2 negative population.

ELIGIBILITY:
Inclusion Criteria - All Patients

* Histologically verified inoperable locally advanced or metastatic adenocarcinoma of the oesophagus, oesophago-gastric junction, or stomach.
* Completion of 18 weeks of first-line chemotherapy with either CX/ CAPOX or FOLFOX (HER2 negative) or CX/ CF + trastuzumab (HER2 positive) for locally advanced / metastatic disease with > stable disease on the end of treatment CT scan (HER2 positive patients must have received at least one cycle of trastuzumab alongside first line chemotherapy; patients receiving chemotherapy delivered on a 3-weekly basis eg CX/ CAPOX should have received 6 cycles and on a two weekly basis e.g. FOLFOX should have received 9 cycles).
* Disease which, following first-line chemotherapy, remains inoperable and unsuitable for definitive chemoradiotherapy.
* Able to proceed with maintenance treatment within 28 days of the last day of the last cycle of chemotherapy.
* Formalin fixed paraffin embedded (FFPE) blocks of diagnostic tissue available for biomarker analysis.
* Any prior chemotherapy or radiotherapy in the adjuvant setting must have been completed at least 6 months prior to the first occurrence of metastatic disease.
* No prior radiotherapy in the advanced disease setting. Patients receiving palliative radiotherapy to sites of disease that are not measurable may be eligible and should be discussed with the Chief Investigator.
* Male/female patients aged ≥18 years.
* WHO Performance status 0, 1 or 2.
* Patients should have a projected life expectancy of at least 3 months.
* Adequate bone marrow function: absolute neutrophil count (ANC) ≥1.5x109/l; white blood cell count ≥ 3x109/l; platelets ≥ 100x109/l; haemoglobin (Hb) ≥ 9g/dl (can be post-transfusion).
* Adequate renal function: calculated creatinine clearance ≥50ml/minute.
* Adequate liver function: serum bilirubin ≤1.5x ULN; aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≤2.5 x ULN (5 × ULN is acceptable for ALT, AST and ALP if liver metastases are present).
* Women of childbearing potential as well as fertile men and their partners must agree to abstain from sexual intercourse or to use an effective form of contraception during the study and for 7 months following the last dose of assigned study drug(s).
* Written informed consent must be obtained from the patient before any study-specific procedures are performed.

Exclusion Criteria - All Patients

* Concurrent enrolment in another clinical trial unless it is an observational (non-interventional) clinical study.
* Tumours of squamous histology.
* Documented brain metastases, central nervous system metastases or leptomeningeal disease.
* Patients who have not recovered from clinically significant effects of any prior surgery, radiotherapy or any other anti-neoplastic therapies. All toxicities must have resolved to grade 1 or less, with the exception of peripheral neuropathy which must be less than or equal to grade 2 according to NCI CTCAE version 4.0.
* Any major surgery within 4 weeks prior to the start of study treatment.
* Uncontrolled hypertension (systolic blood pressure >180 mm Hg or diastolic blood pressure >100 mm Hg).
* Clinically significant (i.e. active) cardiac disease e.g. symptomatic coronary artery disease, symptomatic congestive heart failure, uncontrolled cardiac dysrhythmia, or myocardial infarction within the last 12 months. Patients with any prior history of clinically significant cardiac failure are excluded from study entry.
* History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis) or evidence of interstitial lung disease on baseline chest CT scan.
* Lack of physical integrity of the upper gastro-intestinal tract, malabsorption syndrome, or inability to take oral medication.
* Patients who are pregnant or lactating.
* Known positive tests for human immunodeficiency virus (HIV) infection, hepatitis A or C virus, acute or chronic active hepatitis B infection.
* Other clinically significant disease or co-morbidity which may adversely affect the safe delivery of treatment within this trial.
* Any other malignancies within the last 3 years (other than curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix).
* Treatment with another investigational agent within 30 days of commencing study treatment.

Additional Inclusion / Exclusion Criteria - HER-2 Negative Patients (Arm A)

* Patients must have histologically or cytologically confirmed HER-2 negative disease (HER-2 0-2 by IHC; note if ISH testing is performed this must not demonstrate evidence of gene amplification).
* Patients with known capecitabine intolerance are excluded. This includes patients with previous coronary artery spasm or chest pain deemed to be capecitabine-related.
* Patients with homozygous DPYD gene mutations are excluded. Patients with heterozygous DPYD gene mutations who have tolerated dose-reduced fluoropyrimidines during first-line chemotherapy as per local guidelines are eligible.
* Prior treatment with a PARP inhibitor is excluded (only applicable for A4 & A5 patients).
* Any Grade 3 or 4 GI bleeding within 3 months prior to enrollment are excluded
* Any Grade 3 or 4 venous thromboembolic event (VTE) that is considered by the investigator to be life threatening or that is symptomatic and not adequately treated by anticoagulation therapy, within 3 months prior to randomization are excluded.
* History of GI perforation within 6 months of randomisation are excluded
* History of hepatic encephalopathy or cirrhosis (level Child-Pugh B or worse) are excluded
* Patients must have adequate coagulation function as defined by International Normalised Ratio (INR) ≤1.5 and a partial thromboplastin time/activated partial thromboplastin time (PTT or aPTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy. Patients receiving warfarin must be switched to low molecular weight heparin prior to randomisation.
* Patients with a serious or non-healing wound, ulcer or bone fracture within 28 days prior to randomisation are excluded.
* The patient's urinary protein is ≤1+ on dipstick or routine urinalysis (if urine dipstick is

  * 2+, a 24 hour urine collection for protein must demonstrate < 1000mg of protein in 24 hours.
* Patients experiencing thromboembolic events, including but not limited to myocardial infarction, transient ischaemic attack, cerebrovascular accident, unstable angina, within 6 months prior to first dose of protocol therapy are excluded.
* Patients who have undergone major surgery within 28 days prior to first dose of protocol therapy, or minor surgery/ subcutaneous venous access device placement within 7 days prior to first dose of protocol therapy are excluded.
* Patients receiving chronic anti-platelet therapy or NSAIDS including ibuprofen, naproxen, dipyridamole or clopidogrel, or similar agents are excluded. Once daily aspirin use (up to 325mg/day) is permitted.

Additional Inclusion / Exclusion Criteria - HER-2 Positive Patients (Arm B)

* Patients must have histologically or cytologically confirmed HER-2 positive disease (HER-2 3+ by IHC or HER-2 2+ by IHC and HER-2 gene amplified by ISH).
* Patients must have left ventricular ejection fraction (LVEF) >50% as measured by echocardiogram or >45% measured by MUGA (must also be greater than lower limit of normal at institution).
* Patients with active or prior history of New York Heart Association (NYHA) congestive heart failure are excluded.
* Patients with a known history of hypersensitivity to trastuzumab or any of its components are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2015-02; Primary Completion 2025-04-17 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 5 years
  The progression free survival will be calculated from the date of randomisation to the date of disease progression according to RECIST 1.1 criteria or death from any cause, whichever comes first. In HER 2 negative patients the PFS will be compared between the standard Arm (A1) and capecitabine (A2) and then separately between standard arm (A1) and MEDI 4736 (A3), or standard arm (A1) and Rucaparib (A4), or standard arm (A1) and Ramucirumab (A5).

SECONDARY OUTCOMES:
Progression - free rate (PFR) | 5 years
  Progression-free rate (defined as stable disease, partial or complete response) at 12 weeks (3 months) , 24 weeks (6 months) and 52 weeks (1 year) will be evaluated using RECIST 1.1 criteria. Progression events will be determined by local investigator assessment, and will be collected for up to a 5 year period.
Overall survival (OS) | 5 years
  Will be calculated from the date of randomisation until the date of death from any cause. Patients remaining alive at the time of the analysis will be censored a the date of last follow up.
Objective response rate (ORR) by RECIST 1.1 | 5 years
  This will be evaluated according to RECIST 1.1.
The number of participants with treatment related adverse events as assessed by CTCAE v 4.0 | 5 years
  The number of participants with treatment related adverse events as assessed by CTCAE v 4.0
Analysis of PFS may also be conducted according to biomarker status in relevant arms. For example in HER2 negative patients outcomes in Arm A1 and A3 may be compared according to PDL1 expression status assessed by immunohistochemistry on tissue. | 5 years
  Analysis of PFS may also be conducted according to biomarker status in relevant arms. For example in HER2 negative patients outcomes in Arm A1 and A3 may be compared according to PDL1 expression status assessed by immunohistochemistry on tissue.
Analysis of PFR may also be conducted according to biomarker status in relevant arms. For example in HER2 negative patients outcomes in Arm A1 and A3 will be compared according to PDL1 expression status assessed by immunohistochemistry on tissue. | 5 years
  Analysis of PFR may also be conducted according to biomarker status in relevant arms. For example in HER2 negative patients outcomes in Arm A1 and A3 will be compared according to PDL1 expression status assessed by immunohistochemistry on tissue.
Analysis of OS may also be conducted according to biomarker status in relevant arms. For example in HER2 negative patients outcomes in Arm A1 and A3 will be compared according to PDL1 expression status assessed by immunohistochemistry on tissue. | 5 years
  Analysis of OS may also be conducted according to biomarker status in relevant arms. For example in HER2 negative patients outcomes in Arm A1 and A3 will be compared according to PDL1 expression status assessed by immunohistochemistry on tissue.
Analysis of ORR may also be conducted according to biomarker status in relevant arms. For example in HER2 negative patients outcomes in Arm A1 and A3 will be compared according to PDL1 expression status assessed by immunohistochemistry on tissue. | 5 years
  Analysis of ORR may also be conducted according to biomarker status in relevant arms. For example in HER2 negative patients outcomes in Arm A1 and A3 will be compared according to PDL1 expression status assessed by immunohistochemistry on tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Downs Road, Sutton, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Following trial completion the trial will be submitted for publication to a peer reviewed journal

REFERENCES:
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069